CLINICAL TRIAL: NCT05280093
Title: Hybrid Epicardial and Endocardial Sinus Node Sparing Ablation Therapy for Inappropriate Sinus Tachycardia
Brief Title: HEAL-IST IDE Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-2021-04
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-11

CONDITIONS: Inappropriate Sinus Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Hybrid sinus node sparing ablation procedure (Experimental): Hybrid sinus node sparing ablation procedure using the ISOLATOR Synergy Surgical Ablation System
  Interventions: Device: AtriCure ISOLATOR Synergy Surgical Ablation System

INTERVENTIONS:
Device: AtriCure ISOLATOR Synergy Surgical Ablation System — Hybrid sinus node sparing ablation procedure using the ISOLATOR Synergy Surgical Ablation System

SUMMARY:
Inappropriate Sinus Tachycardia (IST) is a prevalent and debilitating condition in otherwise healthy younger patients, resulting in significant loss of quality of life, lacking effective treatment options or systematic clinical evidence to support a therapy. The primary objective of this clinical trial is to evaluate the safety and effectiveness of a hybrid sinus node sparing ablation procedure for the treatment of symptomatic drug refractory or drug intolerant IST.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years and ≤ 75 years at time of enrollment consent
2. Subject has a diagnosis of IST
3. Documentation of refractoriness (intolerance or failure) of a drug (e.g., rate control drugs such as beta-blockers/calcium channel blockers, ivabradine), and/or AADs
4. Subject is willing and able to provide written informed consent

Exclusion Criteria:

1. Subjects on whom cardiac surgery or single lung ventilation cannot be performed
2. Subjects with indication for or existing ICDs/Pacemakers
3. Presence of channelopathies
4. Previous cardio-thoracic surgery
5. Left Ventricular Ejection Fraction (LVEF) < 50%
6. Body Mass Index (BMI) ≥ 35
7. Presence of supraventricular or ventricular tachycardia
8. Presence of Postural Orthostatic Sinus Tachycardia (POTS)
9. Presence of congenital heart disease
10. History suggestive of secondary cause of tachycardia such as pheochromocytoma, anemia, thyrotoxicosis, chronic fever of unknown origin, COPD, long-term bronchodilators use, severe asthma or carcinoid syndrome
11. Subjects who have had a previous catheter ablation in the right atrium for IST or other disorders
12. Life expectancy < 24 months
13. Pregnant or planning to become pregnant during trial
14. Subjects with substance abuse
15. Subjects with previous weight loss surgery
16. Subject is unwilling and/or unable to return for scheduled follow-up visits
17. Current participation in another clinical investigation of a medical device or a drug, or recent participation in such a trial that may interfere with trial results
18. Not competent to legally represent him or herself (e.g., requires a guardian or caretaker as a legal representative) and;
19. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint | 12-months Post Procedure
  Freedom from IST at 12-months. Freedom from IST is defined as mean heart rate of ≤ 90bpm or at least a 15% reduction in mean heart rate as compared to baseline, in the absence of new or higher dosage of previously failed medications.
Primary Safety Endpoint | 30-days Post Procedure
  Incidence of device or procedure-related major adverse events (MAEs) for subjects undergoing the hybrid sinus node sparing ablation procedure from the index procedure through 30-days post procedure

SECONDARY OUTCOMES:
6-Minute Walk Test | 24-months Post Procedure
  Change in 6-Minute Walk Test (6-MWT) from baseline compared to 6-, 12- and 24-months post-procedure
Borg dyspnea score | 24-months Post Procedure
  Change in Borg dyspnea severity of breathlessness and fatigue score from baseline compared to 6-, 12- and 24-months post-procedure. Borg dyspnea score will be assessed at each of the 6-MWT.
Self-Rating Anxiety Scale | 24-months Post Procedure
  Change from baseline in psychological evaluation compared to 6-, 12- and 24-months post-procedure utilizing the Self-Rating Anxiety Scale (SAS)
IST symptom reduction | 24-months Post Procedure
  IST symptom reduction at baseline to 6-, 12- and 24-months post-procedure
QoL - SF-12 | 24-months Post Procedure
  Change in QoL based on a Short Form Survey (SF-12) domain and component scores at baseline compared to 6-, 12- and 24-months post-procedure
Mean heart rate | 24-months Post Procedure
  Change in mean heart rate at 6-, 12- and 24-months post-procedure compared to baseline, using 7-day continuous monitoring
Reduction in mean heart rate in the absence of rate control drugs | 24-months Post Procedure
  Freedom from IST or at least 15% reduction in mean heart rate at 12- and 24-months compared to baseline, in the absence of rate control drugs (beta-blockers/calcium channel blockers, ivabradine) and/or AADs
Reduction in mean heart rate regardless of rate control drugs | 24-months Post Procedure
  Freedom from IST or at least a 15% reduction in mean heart rate at 12- and 24-months compared to baseline, regardless of rate control drugs (beta-blockers/calcium channel blockers, ivabradine) and/or AADs
Device or procedure related Serious Adverse Events | 12-months Post Procedure
  Device or procedure related Serious Adverse Events (SAEs) through 12-months
Improved heart rate variability - 7-day monitor | 12-months Post Procedure
  Improved heart rate variability for subjects using 7-day continuous monitoring
Improved heart rate variability - Implantable loop recorder | 12-months Post Procedure
  Improved heart rate variability and activity levels for subjects with implantable loop recorders (ILRs)
Health Economics | 24-months Post Procedure
  Health Economics: ER visits and readmissions

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute; Mark La Meir, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Carlo de Asmundis, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Thomas Beaver, MD, Principal Investigator — University of Florida
Locations (26):
- United States (20):
  - Loma Linda University Health, Loma Linda, California
  - Sequoia Hospital, Redwood City, California
  - Stanford University, Redwood City, California
  - Saint Vincent's Medical Center, Bridgeport, Connecticut
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Baptist Health, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - St. Joseph's Hospital / Baycare Health System, Tampa, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Kansas City Cardiac Arrhythmia Research LLC, Overland Park, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - TriHealth, Inc., Cincinnati, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Intermountain Healthcare, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- UZ Brussels, Brussels, Belgium
- San Raffaele Hospital, Milan, Italy
- Netherlands (2):
  - Amsterdam University Medical Center, Amsterdam
  - Maastricht University Medical Center, Maastricht
- Central Clinic Hospital, Warsaw, Poland
- Northern General Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Olshansky B, Sullivan RM. Inappropriate sinus tachycardia. Europace. 2019 Feb 1;21(2):194-207. doi: 10.1093/europace/euy128. PMID 29931244
- [Background] Pellegrini CN, Scheinman MM. Epidemiology and definition of inappropriate sinus tachycardia. J Interv Card Electrophysiol. 2016 Jun;46(1):29-32. doi: 10.1007/s10840-015-0039-8. Epub 2015 Aug 27. PMID 26310298
- [Background] Khiabani AJ, Greenberg JW, Hansalia VH, Schuessler RB, Melby SJ, Damiano RJ Jr. Late Outcomes of Surgical Ablation for Inappropriate Sinus Tachycardia. Ann Thorac Surg. 2019 Oct;108(4):1162-1168. doi: 10.1016/j.athoracsur.2019.03.103. Epub 2019 May 8. PMID 31077661
- [Background] de Asmundis C, Chierchia GB, Sieira J, Stroker E, Umbrain V, Poelaert J, Brugada P, La Meir M. Sinus Node Sparing Novel Hybrid Approach for Treatment of Inappropriate Sinus Tachycardia/Postural Orthostatic Sinus Tachycardia With New Electrophysiological Finding. Am J Cardiol. 2019 Jul 15;124(2):224-232. doi: 10.1016/j.amjcard.2019.04.019. Epub 2019 Apr 23. PMID 31084999
- [Background] Sheldon RS, Grubb BP 2nd, Olshansky B, Shen WK, Calkins H, Brignole M, Raj SR, Krahn AD, Morillo CA, Stewart JM, Sutton R, Sandroni P, Friday KJ, Hachul DT, Cohen MI, Lau DH, Mayuga KA, Moak JP, Sandhu RK, Kanjwal K. 2015 heart rhythm society expert consensus statement on the diagnosis and treatment of postural tachycardia syndrome, inappropriate sinus tachycardia, and vasovagal syncope. Heart Rhythm. 2015 Jun;12(6):e41-63. doi: 10.1016/j.hrthm.2015.03.029. Epub 2015 May 14. No abstract available. PMID 25980576
- [Background] Nwazue VC, Paranjape SY, Black BK, Biaggioni I, Diedrich A, Dupont WD, Robertson D, Raj SR. Postural tachycardia syndrome and inappropriate sinus tachycardia: role of autonomic modulation and sinus node automaticity. J Am Heart Assoc. 2014 Apr 10;3(2):e000700. doi: 10.1161/JAHA.113.000700. PMID 24721800
- [Background] Masumoto A, Takemoto M, Mito T, Tanaka A, Kawano Y, Kumeda H, Kang H, Matsuo A, Hida S, Okazaki T, Tayama KI, Yoshitake K, Kosuga K. Inappropriate Sinus Tachycardia Diagnosed and Treated as Depression Successfully Treated by Radiofrequency Catheter Ablation. Intern Med. 2017;56(5):523-526. doi: 10.2169/internalmedicine.56.7579. Epub 2017 Mar 1. PMID 28250298
- [Background] Yasin OZ, Vaidya VR, Chacko SR, Asirvatham SJ. Inappropriate Sinus Tachycardia: Current Challenges and Future Directions. J Innov Card Rhythm Manag. 2018 Jul 15;9(7):3239-3243. doi: 10.19102/icrm.2018.090706. eCollection 2018 Jul. No abstract available. PMID 32479576
- [Background] Cappato R, Castelvecchio S, Ricci C, Bianco E, Vitali-Serdoz L, Gnecchi-Ruscone T, Pittalis M, De Ambroggi L, Baruscotti M, Gaeta M, Furlanello F, Di Francesco D, Lupo PP. Clinical efficacy of ivabradine in patients with inappropriate sinus tachycardia: a prospective, randomized, placebo-controlled, double-blind, crossover evaluation. J Am Coll Cardiol. 2012 Oct 9;60(15):1323-9. doi: 10.1016/j.jacc.2012.06.031. Epub 2012 Sep 12. PMID 22981555
- [Background] Kreisel D, Bailey M, Lindsay BD, Damiano RJ Jr. A minimally invasive surgical treatment for inappropriate sinus tachycardia. J Thorac Cardiovasc Surg. 2005 Aug;130(2):598-9. doi: 10.1016/j.jtcvs.2004.12.026. No abstract available. PMID 16077449
- [Background] de Asmundis C, Chierchia GB, Lakkireddy D, Romeya A, Okum E, Gandhi G, Sieira J, Vloka M, Jones SD, Shah H, Winner M, Patel D, Whalen SP, Beaty EH, Kincaid EH, Lee A, Brodt C, Taylor BJ, Colombowala I, Romano M, Morady F, Stroker E, Overeinder I, Bala G, Van Meeteren J, Krauthammer Y, Koerber S, Shults C, Thomaides A, Badhwar N, Gopinathannair R, Shah A, Tummala R, Bello D, Hoff S, Almorad A, Frazier K, Brugada P, La Meir M. Sinus node sparing novel hybrid approach for treatment of inappropriate sinus tachycardia/postural sinus tachycardia: multicenter experience. J Interv Card Electrophysiol. 2022 Apr;63(3):531-544. doi: 10.1007/s10840-021-01044-5. Epub 2021 Aug 23. PMID 34424446
- [Background] C. De Asmundis et al, "Thoracoscopic Ablation of Inappropriate Sinus Tachycardia and Postural Orthostatic Tachycardia Syndrome." Hands-On-Ablation, The Expert's Approach, Third Edition.
- [Background] Lakkireddy D, Garg J, DeAsmundis C, LaMeier M, Romeya A, Vanmeetren J, Park P, Tummala R, Koerber S, Vasamreddy C, Shah A, Shivamurthy P, Frazier K, Awasthi Y, Chierchia GB, Atkins D, Bommana S, Di Biase L, Al-Ahmad A, Natale A, Gopinathannair R. Sinus Node Sparing Hybrid Thoracoscopic Ablation Outcomes in Patients with Inappropriate Sinus Tachycardia (SUSRUTA-IST) Registry. Heart Rhythm. 2022 Jan;19(1):30-38. doi: 10.1016/j.hrthm.2021.07.010. Epub 2021 Jul 30. PMID 34339847
- [Background] Calkins H, Hindricks G, Cappato R, Kim YH, Saad EB, Aguinaga L, Akar JG, Badhwar V, Brugada J, Camm J, Chen PS, Chen SA, Chung MK, Nielsen JC, Curtis AB, Davies DW, Day JD, d'Avila A, de Groot NMSN, Di Biase L, Duytschaever M, Edgerton JR, Ellenbogen KA, Ellinor PT, Ernst S, Fenelon G, Gerstenfeld EP, Haines DE, Haissaguerre M, Helm RH, Hylek E, Jackman WM, Jalife J, Kalman JM, Kautzner J, Kottkamp H, Kuck KH, Kumagai K, Lee R, Lewalter T, Lindsay BD, Macle L, Mansour M, Marchlinski FE, Michaud GF, Nakagawa H, Natale A, Nattel S, Okumura K, Packer D, Pokushalov E, Reynolds MR, Sanders P, Scanavacca M, Schilling R, Tondo C, Tsao HM, Verma A, Wilber DJ, Yamane T. 2017 HRS/EHRA/ECAS/APHRS/SOLAECE expert consensus statement on catheter and surgical ablation of atrial fibrillation. Heart Rhythm. 2017 Oct;14(10):e275-e444. doi: 10.1016/j.hrthm.2017.05.012. Epub 2017 May 12. No abstract available. PMID 28506916
- [Background] Broglio KR, Connor JT, Berry SM. Not too big, not too small: a goldilocks approach to sample size selection. J Biopharm Stat. 2014;24(3):685-705. doi: 10.1080/10543406.2014.888569. PMID 24697532